CLINICAL TRIAL: NCT01376440
Title: Acceptability and Effectiveness of Household Water Chlorination in Reducing the Prevalence of Diarrhea Among Under Five Children in Eastern Ethiopia
Brief Title: Acceptability and Effectiveness of Household Water Treatment in Reducing Diarrhea Among Under Five Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haramaya Unversity (Other)
Responsible Party: Principal Investigator, Bezatu Mengiste, Mr, Haramaya Unversity
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SGS13/15/11
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Acute Diarrhoea
Keywords: three or more loss stools in 24 hours
MeSH Terms: interventions — Sodium Hypochlorite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Household water treatment (Experimental): household water treatment with 1.25% sodium hypochlorite
  Interventions: Other: household water treatment
- control (No Intervention): Usual practice (the use of "Jerrican" for water storage, which is considered as safe storage)

INTERVENTIONS:
Other: household water treatment — household water treatment with 1.25% sodium hypochlorite
  Other Names: 1.25% sodium hypochlorite
  Arms: Household water treatment

SUMMARY:
The Millenium development goals (MDGs) call for reducing by half the proportion of people without sustainable access to safe drinking water. This goal was adopted in large part because safe drinking water has been seen as critical to fighting diarrheal disease. Source protection is considered the main intervention area to achieve this goal. However, research worldwide that has shown that even drinking water which is safe at the source is subject to frequent and extensive fecal contamination during collection, storage and use in the home. This contamination is through the introduction of cups, dippers or hands, contamination by flies, cockroaches, and rats. Even piped water supplies of adequate microbial quality can pose infectious disease risks if they become contaminated due to unsanitary collection, storage conditions and practices within households.

To reduce this problem, point-of-use water treatment has been advocated as a means to substantially decrease the global burden of diarrhea and to contribute to the MDGs. However, research indicates that there are many unanswered questions around Household water treatment (HWT) that require small or medium scale epidemiological studies and randomized controlled trials, especially with regard to effectiveness, acceptability and identifying suitable target populations. Some of the most urgent questions to be resolved are:(1) How much of the currently cited disease reduction of HWT is due to bias? (2) What is the effect of HWT on nutritional status (weight gain and growth)?(3) At which populations should HWT be targeted? (4) Is it acceptable and sustainable in poor communities where the risk of diarrheal disease is high.

hypothesis: Do household water treatment with chlorine reduce diarrhea among underfive children? hypothesis: Do household water treatment with chlorine acceptable in the community?

ELIGIBILITY:
Inclusion Criteria:

* All children under five years of age in the randomly selected clusters of Kersa district

Exclusion Criteria:

* seriously sick children in the randomly selected clusters of Kersa district

Ages: 1 Month to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 845 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To assess the prevalence of diarrhea among under five children | four months
  weekly visit of the household for the presence of diarrhoea among underfive for four months in both the intervention and control groups

SECONDARY OUTCOMES:
To assess the weight gain among the intervention and control groups of under five children | At the beginning and end of the study ( 4 months interval)
  This is designed to assess whether there is weight gain (objective outcome) in children assigned to the intervention group compared to the control group. It is supplement to the prevalence of diarrhea which is subjective outcome for this study
Residual chlorine test | four months
  The use of the intervention (1.25% hypochlorite) is confirmed by the testing the residual chlorine weekly for for months from each household assigned in the intrevention group

CONTACTS AND LOCATIONS:
Overall Officials: Bezatu M Alemu, M.Sc, Principal Investigator — Assistant professor
Locations (1):
- Kersa district, Kersa, Eastern Hararage, Ethiopia

REFERENCES:
- [Derived] Mengistie B, Berhane Y, Worku A. Household water chlorination reduces incidence of diarrhea among under-five children in rural Ethiopia: a cluster randomized controlled trial. PLoS One. 2013 Oct 23;8(10):e77887. doi: 10.1371/journal.pone.0077887. eCollection 2013. PMID 24194899